CLINICAL TRIAL: NCT05925465
Title: Effect of Combined Maxillary and Mandibular Nerve Block on Orthognathic Surgery Outcomes
Brief Title: Maxillary and Mandibular Nerve Block
Acronym: nerve block
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Assistant Professor of Anesthesia and Surgical Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Jaw nerve block
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of two groups, each of 30 patients, by means of coded envelopes to receive bilateral combined maxillary and mandibular nerve block (MNB group) or not receive any nerve block (control group)
Who Masked: Participant, Investigator
Masking Description: Nerve block will be done by an anesthesiologist who will not be involved in data collection to ensure blindness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maxillary and mandibular nerve block (MMNB) group (Active Comparator): receive bilateral combined maxillary and mandibular nerve block. Three mL of 0.5% isobaric bupivacaine will be injected for each nerve block after negative aspiration of blood.
  Interventions: Procedure: Maxillary and mandibular nerve block
- Control (C) group (Placebo Comparator): not receive any nerve block
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Maxillary and mandibular nerve block — receive bilateral combined maxillary and mandibular nerve block
  Arms: Maxillary and mandibular nerve block (MMNB) group
Other: Control — not receive any nerve block
  Arms: Control (C) group

SUMMARY:
Mandibular fractures are among the most common (60-70%) maxillofacial fractures observed in emergency rooms. In the closed reduction (non-surgical), the bone fragments are realigned manually or by using traction devices. The open reduction surgery of mandibular fractures should first ensure the restoration of the occlusion of the mandible to prevent postoperative malocclusion, followed by stabilization by means of rigid fixations such as plates, screws, and rigid intermaxillary blocks in order to minimise any nonunion, malunion, or delayed union of the fracture segments. These surgical procedures are associated with moderate postoperative pain, being the first 24 hours the most intense pain period. Maxillary and mandibular nerve blocks are performed in patients with refractory trigeminal neuralgia. However, there have been few studies evaluating the analgesic effects of these blocks for maxillofacial surgeries.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I/II patients,
* within the age group of 21-60 years
* both sex
* scheduled for elective faciomaxillary surgery

Exclusion Criteria:

* Pregnant or breast-feeding women
* Patients with polytrauma
* Patients necessitating postoperative ventilation
* Oral or facial infection
* Coagulopathy
* Drug intake for chronic pain
* Known allergy to the study drugs
* Psychiatric disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Total postoperative fentanyl rescue analgesic consumption | first 24 hours postoperatively
  microgram

SECONDARY OUTCOMES:
Intraoperative heart rate (HR) | each 15 minutes Intraoperative plus 1hour postoperatively and 2hours postoperatively
  beats per minute
Intraoperative mean arterial pressure (MAP) | each 15 minutes Intraoperative plus 1hour postoperatively and 2hours postoperatively
  mmHg
10-cm visual analogue scale (VAS) | at 0, 2, 4, 6, 8, 12, and 24 hours postoperatively
  where 0 represented no pain, and 10 meant the worst possible pain
Postoperative analgesic duration | up to 24 hours (the time from ending of the nerve block till the first rescue morphine dose)
  hours
Patients' satisfaction about their analgesia | 24 hours postoperatively
  on a scale from 1 (poor), 2 (fair) to 3 (good)
Total postoperative diclofenac sodium consumption | 24 hours postoperatively
  mg
The total Intraoperative supplementary fentanyl | during the intraoperative duration
  microgram

CONTACTS AND LOCATIONS:
Locations (1):
- Maha Ahmed AboZeid, Al Mansurah, Mansoura, Egypt

IPD SHARING:
Plan to Share IPD: No